CLINICAL TRIAL: NCT02865629
Title: N-acetylcysteine in the Treatment of Depressive Symptoms in Youth at High-risk for Bipolar Disorder: a Functional Connectivity Study
Brief Title: N-acetylcysteine in the Treatment of Depressive Symptoms in Bipolar Offspring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Fabiano Nery, Assistant Professor of Psychiatry in the Department of Psychiatry and Behavioral Neuroscience, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nery UCNI NAC study
Record Dates: First submitted 2016-06-28; First posted 2016-08-12 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-acetyl cysteine (Experimental): Following the screening and review of all laboratory studies, patients will be scheduled to receive N-acetylcysteine.
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — N-acetylcysteine will be initiated at 600 mg PO daily for Week 1, then increased to 600 mg PO twice a day for Week 2, then increased to 600 mg PO morning and 1200 mg PO evening for Week 3, and then increased to 1200 mg PO twice a day for Week 4-8. Doses might be decreased anytime if clinically indicated. Following the study, all patients will be referred to treatment as usual. Adherence will be assessed in weekly visits in the first month and then bi-weekly in the second month. Adherence will be assessed by subject interview, pill counts during each study visit, and by legal guardian interview (if minor).
  Other Names: Acetylcysteine

SUMMARY:
N-acetylcysteine in the treatment of depressive symptoms in youth at high-risk for bipolar disorder: a functional connectivity study

DETAILED DESCRIPTION:
To conduct an 8-week, open label study of N-acetylcysteine for the treatment of depressive symptoms in youth at high risk for bipolar disorder, with resting state functional magnetic resonance imaging (fMRI) examinations at baseline and endpoint. This proposal is innovative because it investigates the efficacy and tolerability of a novel pharmacological treatment in youth offspring of bipolar disorder, and examines the neurophysiology of predictors of mood disorders in youth at high risk for bipolar disorder. This study will obtain pilot data to propose a larger, neuroimaging-based, double-blind, placebo-controlled trial of N-acetylcysteine in youth at high risk for bipolar disorder. The expected outcome, that N-acetylcysteine will be efficacious in ameliorating depressive symptoms in youth at high risk for bipolar disorder, and that it will demonstrate improvement in functional connectivity within the left frontostriatal circuit associated with treatment response.

ELIGIBILITY:
Inclusion:

1. Male or female subjects 15 years, 0 months - 24 years, 11 months of age at screening
2. For minor, at least one parent or step-parent/guardian with whom the subject lives is willing to participate in research sessions
3. For minor, the child and relative(s) are able and willing to give written informed assent/consent to participate, respectively
4. Subject has at least one first degree relative with Bipolar I Disorder, as assessed by the Structured Clinical Interview for DSM (SCID) or the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS-PL)
5. Subject shows evidence of current significant depressive symptoms as determined by a current Hamilton Depression Rating Scale (HAM-D) greater or equal to 8

Exclusion:

1. Patient has presence of current or lifetime history of manic or hypomanic mood episodes, psychotic disorders including schizophrenia, current major depressive episode, and/or more than two prior major depressive episodes
2. Patient has a DSM-5 diagnosis of autism, pervasive developmental disorder, OCD, PTSD, or Tourette's disorder
3. Patient has drug or alcohol abuse or dependence disorders in the three months prior to study recruitment, although a lifetime history of substance or alcohol disorders can be present if the patient has been abstinent for at least three months
4. Pregnancy; participants will be encouraged but not mandated to discuss a positive pregnancy test with their guardians (if minors) and we will follow local laws
5. Patient has history of major neurological disorders (such as epilepsy), or head trauma with > 10 minutes loss of consciousness
6. Patient has evidence of mental retardation (IQ less than 70), as determined by the Wechsler Abbreviated Scale of Intelligence (WASI)
7. Patient has any contraindication for MRI, including metal in the body related to an injury or surgery (e.g., surgical clips, metal fragments in the eyes), piercings that cannot be removed, or braces
8. Patient has history of allergic reaction to N-acetylcysteine

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) scores | Baseline to endpoint (8 weeks)
  The primary outcome will be change in depressive symptoms, as measured by HAMD scores, from baseline to endpoint.

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS) scores | Baseline to endpoint (8 weeks)
  A secondary outcome will be change in manic symptom, measured by YMRS scores, from baseline to endpoint.
Hamilton Anxiety Rating Scale (HAM-A) scores to measure anxiety symptoms | Baseline to endpoint (8 weeks)
  A secondary outcome will be change anxiety symptoms, as measured by HAM-A scores, from baseline to endpoint.
Clinical Global Impression of Severity (CGI-S) scores | Baseline to endpoint (8 weeks)
  A secondary outcome will be change in subjects' overall clinical condition, as measured by CGI-S scores, from baseline to endpoint.
Connectivity index, as defined by the temporal bivariate correlation between fMRI signal fluctuations in the left ventrolateral prefrontal cortex and the left striatum | Baseline to endpoint (8 weeks)
  A secondary outcome will be change in functional connectivity, as measured by the connectivity index, between the left ventrolateral prefrontal cortex and the left striatum from baseline to endpoint. The connectivity index is defined as the temporal bivariate correlation between fMRI signal fluctuations in the 2 regions of interest.
Correlation between change in depressive symptoms and change in connectivity index | Baseline to endpoint (8 weeks)
  A secondary outcome will be correlation between changes in depressive symptoms and changes in functional connectivity, as measured by the connectivity index, between the left ventrolateral prefrontal cortex and left striatum from baseline to endpoint. The connectivity index is defined as the temporal bivariate correlations between fMRI signal fluctuations in the 2 regions of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiano G. Nery, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Department of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No